CLINICAL TRIAL: NCT00594256
Title: Open Label, Pilot Study of Adjunctive Xyrem (Sodium Oxybate) for the Treatment of Schizophrenia and Associated Sleep Disturbances
Brief Title: Sodium Oxybate in Schizophrenia With Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Daniel C. Javitt, MD, PhD, Director, Schizophrenia Research Center, Nathan Kline Institute for Psychiatric Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07I/C36-0
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Schizophrenia; Insomnia Related to Schizophrenia (307.42)
Keywords: Schizophrenia; Sleep Architecture; Sodium Oxybate; Insomnia; Cognition
MeSH Terms: conditions — Schizophrenia; Sleep Initiation and Maintenance Disorders | interventions — Sodium Oxybate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sodium oxybate (Experimental): Active treatment
  Interventions: Drug: Sodium Oxybate

INTERVENTIONS:
Drug: Sodium Oxybate — Patients will undergo a one-week evaluation period, which will include a taper and discontinuation of any currently prescribed sedative/hypnotics, as well as baseline diagnostic, psychopathology, neurocognitive and polysomnographic measurements (see below for details). Hypnotic taper may be extended or abbreviated, depending on clinical judgment. Patients will then begin a 4-week trial of adjunctive Xyrem (sodium oxybate). Patients will begin at 4.5 g/night (in divided doses of 2.25 g, with 1st dose at bedtime and then 2nd dose four hours later). Dosage will increase by 1.5 g/day every week, until a dose of 9 g nightly is reached, or a patient cannot tolerate further dose escalations. Medication will be administered in divided dosage for the duration of the study. A three-week taper (by 3 g/day weekly) of sodium oxybate will follow the four-week trial of sodium oxybate.
  Other Names: Xyrem

SUMMARY:
The present protocol proposes study of the recently approved compound sodium oxybate (Xyrem), a gamma-aminobutyric acid type b (GABAB) and a g-hydroxybutyric acid (GHB) receptor agonist, for the study of persistent symptoms of schizophrenia. Sodium oxybate is a central nervous system depressant currently approved for treatment of narcolepsy associated with cataplexy and excessive daytime sleepiness. In addition to evaluating effects on sodium oxybate on persistent symptoms and neurocognitive deficits in schizophrenia, the study will test the hypothesis that this medication may be particularly effective in combating Insomnia Related to Schizophrenia, and in normalizing symptomatic and polysomnographic manifestations of sleep-related brain dysfunction in schizophrenia.

DETAILED DESCRIPTION:
Rationale/Study Hypothesis:

Rationale for study of sodium oxybate is twofold: first, sleep dysfunction is an important and overlooked aspect of schizophrenia intrinsically linked to cognitive and functional impairments, and, second, GABAB receptors regulate dopaminergic and glutamatergic systems in vivo, suggesting that GABAB agonists may be therapeutically beneficial in schizophrenia.

We are aware of three previous trials of GHB in schizophrenia, two of which did not show any overall benefit in psychopathology. We noted multiple limitations in the controlled trials, including:

1. requirement of cumbersome dosing patterns (up to six times a day) that could have led to incomplete compliance,
2. lack of objective measures of subjective sleep or sleep architecture,
3. lack of objective cognitive testing,
4. use of GHB as monotherapy or only in conjunction with only low dose antipsychotics,
5. short trial duration (less than 4 weeks),
6. relatively low overall night-time dose of GHB, and
7. a heterogeneous, small sample.

We propose an open label, proof of concept study evaluating the effect of sodium oxybate on insomnia in schizophrenia. The primary hypothesis of the study is that patients treated with sodium oxybate will show improved subjective sleep as measured by the overall Epworth Sleepiness Scale and the Pittsburgh Sleep Quality Index. Secondarily, we expect superior reduction in total psychopathology and PANSS factor scales (PANSS), polysomnographic measures, and neurocognition (MATRICS).

Design and dosage schedule:

We plan to enroll eight hospitalized patients with diagnostic & statistical manual text revision (DSM-IV-TR) schizophrenia and insomnia related to schizophrenia. The study will include: a one-week evaluation period, which will include tapering of any hypnotics, baseline diagnostic, psychopathology, neurocognitive, electrophysiological and polysomnographic measurements. Patients will then begin a four-week trial of adjunctive sodium oxybate, with a three-week taper of sodium oxybate to follow. Hypnotic/sodium oxybate taper may be extended or abbreviated, depending on clinical judgment.

Patients entering the study will be permitted to receive both typical and atypical antipsychotics. Treating psychiatrists will be encouraged to maintain fixed doses of all psychotropic medication throughout the study.

Other than haloperidol and benztropine prn (up to 10 mg/day of haloperidol), the prescription of a new psychotropic will not be permitted. After the second week of study medication, any subject requiring more than 4 doses of haloperidol in one week will be considered to have relapsed, and will be withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-45 with a DSM-IV diagnosis of schizophrenia and insomnia related to schizophrenia, confirmed by a structured interview (SCID).

Exclusion Criteria:

* Lack of capacity to give informed consent (capacity is determined by a licensed member of the treatment team).
* Unstable medical illness.
* Diagnosis of restless leg syndrome, a seizure disorder, uncontrolled hypertension, unstable cardiac illness, or obstructive sleep apnea.
* Pregnancy or lack of adequate birth control.
* History of substance dependence disorder.
* Current treatment with valproic acid.
* Succinic semialdehyde dehydrogenase deficiency (SSADH).
* Persistent need for treatment with benzodiazepines, barbiturates, opiates or other sedative hypnotics.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Javitt, MD PhD, Principal Investigator — Nathan Kline Institute for Psychiatric Research
Locations (1):
- Nathan Kline Insitute for Psychiatric Research, Orangeburg, New York, United States

REFERENCES:
- [Result] Kantrowitz JT, Oakman E, Bickel S, Citrome L, Spielman A, Silipo G, Battaglia J, Javitt DC. The importance of a good night's sleep: an open-label trial of the sodium salt of gamma-hydroxybutyric acid in insomnia associated with schizophrenia. Schizophr Res. 2010 Jul;120(1-3):225-6. doi: 10.1016/j.schres.2010.03.035. No abstract available. PMID 20435443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Rockland Psychiatric Center
Groups:
- Sodium Oxybate (Open Label): open label sodium oxybate treatment, beginning at 4.5 g/night and increasing weekly to a final dose of 9 g/night. Given in divided dose, half at bedtime and half 4 hours later (subjects were woken up)
Period: Overall Study
Arm/Group | Sodium Oxybate (Open Label)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sodium Oxybate (Open Label)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Pittsburgh Sleep Quality Index
Description: This rating scale generates a global sleep-quality score, as well as scores on 7 components of sleep quality: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The 19 items are combined to form seven "component" scores, each of which has a range of O-3 points. The seven component scores are then added to yield one "global" score, with a range of O-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas.
Time Frame: 1 month
Population: ITT
Measure: Mean (Standard Deviation); unit: global score
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 8
global score | 6.1 (3.7)
Statistical Analysis 1: Comparison: Sodium Oxybate; Open label baseline final paired t test; Test type: Superiority or Other; p = 0.002, t-test, 2 sided

2. Primary Outcome: Epworth Sleepiness Scale
Description: Designed to measure daytime sleepiness. 8 items rated 0-3, with higher scores associated with a greater daytime sleepiness. overall score rated 0-24, with scores greater than 10 indicating significant daytime sleepiness.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: global score
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 8
global score | 4.8 (4.6)
Statistical Analysis 1: Comparison: Sodium Oxybate; Open label baseline final paired t test; Test type: Superiority or Other; p = 0.02, t-test, 2 sided

3. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) Negative Factor
Description: The PANSS Negative factor is a 7-item rating scale widely used in the assessment of schizophrenia. Range is 7-49 with higher scores worse
Time Frame: 1 month
Population: Paired t test of baseline and final values
Measure: Mean (Standard Deviation); unit: mean decrease in negative subscale
Arm/Group | Sodiumn Oxybate
Number analyzed (Participants) | 8
mean decrease in negative subscale | 2.8 (3.2)
Statistical Analysis 1: Comparison: Sodiumn Oxybate; Open label baseline final paired t test; Test type: Superiority or Other; p = 0.04, t-test, 2 sided

4. Secondary Outcome: MATRICS Neurocognitive Battery Composite
Description: This is a series of neurocognitive tests developed by the National Institute of Mental Health to evaluate medications targeting cognition in an efficient and reliable manner. It will be modified by the deletion of the social competence domain. The six domains include speed of processing, attention/vigilance, working memory, verbal learning, visual learning and reasoning/problem solving. The primary outcome will be the mean T-score (mean of six domains).
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: Composite T-score
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 8
Composite T-score | -.26 (3.8)
Statistical Analysis 1: Comparison: Sodium Oxybate; Open label baseline final paired t test; Test type: Superiority or Other; p = 0.8, t-test, 2 sided

5. Secondary Outcome: Slow Wave Sleep Minutes
Description: Overnight sleep study: Subjects will undergo polysomnography four times during this study, on consecutive nights during the observation week and on consecutive nights at the end. Polysomnography will be performed in a modified seclusion room on the in patient unit. The first of the consecutive nights will be used for adaptation to the study conditions. Sleep was recorded between lights off (10 pm) and lights on (at 6:45 am). We aim for conditions for falling asleep as comfortable as possible under the experimental condition.
Time Frame: 1 month
Population: 4 pre post
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sodium Oxybate
Number analyzed (Participants) | 4
minutes | 34.1 (26.0)
Statistical Analysis 1: Comparison: Sodium Oxybate; Open label baseline final paired t test; Test type: Superiority or Other; p < 0.01, t-test, 1 sided

ADVERSE EVENTS:
Arm/Group | Sodium Oxybate (Open Label)
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 5/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Oxybate (Open Label) (N=8)
nausea (Gastrointestinal disorders) | 2 (2)
nocturnal enuresis (Renal and urinary disorders) | 2 (2)
agitation (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Open Label Small sample

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No